CLINICAL TRIAL: NCT02989766
Title: Preparing Mothers for Feeding Their Newborns: A Self-Guided Program for Pregnant Women
Brief Title: A Self-Guided Breastfeeding Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jaye Shyken, MD, MD, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25115
Record Dates: First submitted 2016-10-18; First posted 2016-12-12 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - Intervention (Active Comparator): Education on Breast Feeding 3 activity sheets prenatally-study related. Complete a pre-questionnaire, a pre-delivery and a postpartum questionnaire
  Interventions: Behavioral: Education on Breast Feeding
- B - Standard of Care (No Intervention): Complete a pre-questionnaire, a pre-delivery and a postpartum questionnaire

INTERVENTIONS:
Behavioral: Education on Breast Feeding — Subjects in the intervention arm will complete 3 activity sheets prenatally-study related.
  Arms: A - Intervention

SUMMARY:
This intervention would be a series of self-help-style educational and motivational activity sheets for patients to complete independently. This will be a randomized clinical control trial.

Subjects will complete a pre delivery questionnaire and a postpartum questionnaire. Subjects in the intervention arm will complete 3 activity sheets prenatally during their wait time at the clinic. The first worksheet can be completed the day of recruitment after consent is signed.

Subjects will be contacted by phone at 3 and 6 months postpartum to assess long term duration of breast feeding.

DETAILED DESCRIPTION:
As the benefits of human milk become evident, the investigators are striving to improve the breastfeeding (BF) rate among new mothers. In April and May of 2014, 73 (71%) of well babies received human milk at discharge from our postpartum unit, with 40 (35%) and receiving human milk exclusively. In the neonatal intensive care unit, 83 (89%) received human milk during those months.

Many of the patients at the teaching institution share risk factors for failure to BF, including poverty, obesity, unplanned pregnancy and being African American. Efforts have had limited effect in improving initiation and duration among these patients.

Studies examining the efficacy of various modalities of antenatal education produced modest results in improving initiation and duration of BF. Several studies examined group BF education versus routine prenatal care without significant differences in initiation, exclusivity (the practice of using human milk exclusively and not supplementing with formula) or duration. Conversely, other study showed a difference in initiation with group education and showed a difference in exclusivity. Formalized education compared to routine clinical practice education did not result in a difference in exclusivity in several studies and neither did a program that included a video showed a difference in initiation with formal education.

A few studies compared peer counseling to routine prenatal care. One small study of 59 women found an increase in initiation rate, while a larger study of 2511 women did not find a difference in initiation or duration.

Other studies found no significant difference in initiation, duration or exclusivity with an educational program on practical BF skills nor a program on BF attitudes. A small study that paired BF education with material incentives increased exclusivity. Three studies comparing interventions by lactation consultants found no difference in initiation or duration, although one study showed improvement in exclusivity. Postpartum BF self-efficacy correlates with BF duration and two studies showed improvement in exclusivity with a BF class based on principles of self-efficacy. These studies based their intervention on Bandura's theory of self-efficacy, which proposes that an individual's expectation of personal efficacy will determine her initiation of coping behavior, effort expenditure and duration of persistence. This theory recognizes four components that contribute to an individual's sense of self- efficacy, and these include performance accomplishment, vicarious, or social, experience, verbal persuasion and psychological state. developed a validated scale at measuring prenatal maternal self-efficacy in breastfeeding.

These two studies used a teaching approach that assumes that pregnant women are adults who are self-motivated and have past experience that shapes their learning and are a component to their perception of self-efficacy.

Printed self-help materials are appealing as a low cost intervention that could be widely implemented. Furthermore, a large study among pregnant women showed that a self-help guide that is particularly tailored towards pregnant women could be effective in promoting another healthy behavior modification: smoking cessation. Potentially this method could be effective when used to prepare mothers for breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients < 32 weeks gestation.

Exclusion Criteria:

* Patient who have not had an ultrasound confirming viable intrauterine pregnancy.
* Patients beyond 32 weeks gestation will be excluded as some are unlikely to return for a sufficient number of prenatal visits to complete the intervention.
* Patients with medical contraindications to breastfeeding such as HIV or active substance abuse.
* Patients planning to take medications in the postpartum period that are incompatible with breastfeeding such as anti-metabolites.
* Patients giving birth to a nonviable infant.
* Patients without adequate reading and writing skills to complete the questionnaires and activity sheets.

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 335 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
improving duration of BF. | 16 Months
  It was propose using a 3-part prenatal self-help guide to educate and prepare mothers for breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Jaye Shyken, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No